CLINICAL TRIAL: NCT06540859
Title: Spinal Cord Stimulation for Autonomic Recovery in Inpatient Rehabilitation After Acute SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Soshi Samejima, Assistant Professor: Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00020243
Record Dates: First submitted 2024-06-27; First posted 2024-08-06 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries
Keywords: Transcutaneous Spinal Cord Stimulation; Inpatient Rehabilitation; Cardiovascular Recovery following SCI; Bladder and Bowel Recovery following SCI
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: randomized, single-blind, two-arm sham-controlled clinical trial with two arms (tSCS compared to sham-stimulation) and two parts (Part A and Part B). Part A will be conducted while participants are staying in inpatient rehabilitation. Participants will be randomized to either tSCS or sham stimulation. Part B will take place in outpatient rehabilitation medicine and all participants will receive tSCS stimulation for up to 18 sessions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transcutaneous Spinal Cord Stimulation (Experimental): Device: Transcutaneous Spinal Stimulation
  Non-invasive electrical stimulation of the spinal cord over the skin. A portable tSCS device, SCONE or TESCoN (SpineX Inc., USA), whichever available, will be used to deliver 1ms pulses with 10kHz carrier frequency at 30 Hz, which has demonstrated autonomic recovery in our previous studies. The location of tSCS is predetermined (at T10 and T11 vertebral levels). The stimulation intensity will range from 10 to 200 mA
  Interventions: Device: Transcutaneous Spinal Cord Stimulation
- Sham stimulation (Sham Comparator): Device: Sham Stimulation
  Non-invasive electrical stimulation of a lower extremity muscle group over the skin. The intensity of electrical stimulation will be briefly ramped up to a level at which the participants report perceiving the stimulation (i.e., sensory threshold), then ramped down and turned off for the remainder of the intervention.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation; Device: Sham Stimulation

INTERVENTIONS:
Device: Transcutaneous Spinal Cord Stimulation — Non-invasive electrical stimulation of the spinal cord over the skin. A portable tSCS device, SCONE or TESCoN (SpineX Inc., USA), whichever available, will be used to deliver 1ms pulses with 10kHz carrier frequency at 30 Hz, which has demonstrated autonomic recovery in our previous studies. The location of tSCS is predetermined (at T10 and T11 vertebral levels). The stimulation intensity will range from 10 to 200 mA and specific criteria will be followed to determine the optimal therapeutic stimulation.
  Other Names: tSCS
Device: Sham Stimulation — Non-invasive electrical stimulation of a lower extremity muscle group over the skin. A portable tSCS device, SCONE or TESCoN (SpineX Inc., USA), whichever available, will be used to deliver sham stimulation. The intensity of electrical stimulation will be briefly ramped up to a level at which the participants report perceiving the stimulation (i.e., sensory threshold), then ramped down and turned off for the remainder of the intervention.
  Arms: Sham stimulation

SUMMARY:
This study is a randomized, single-blind, two-arm sham-controlled clinical trial to evaluate the safety and efficacy of transcutaneous spinal cord stimulation (tSCS) over the lower thoracic and upper lumbar spinal cord segments for cardiovascular function in adults (21-65 years old) with cervical and upper thoracic spinal cord injury (SCI) (≥T6) AIS A-D during inpatient rehabilitation and outpatient visits within three months after the onset. We will recruit 26 individuals with SCI, admitted to inpatient rehabilitation facilities (IRFs) or after discharged from IRFs. We will also examine the effect of tSCS on lower urinary tract (LUT) and bowel functions as secondary outcomes.

The main questions this study aims to answer are:

1. Assess the safety of single and repeated tSCS session(s) on cardiovascular function in the acute SCI: We will test the safety of single tSCS at T10-L2 session at rest and during orthostatic challenge (i.e., situ-up tests) at the baseline and the effect of five tSCS sessions on cardiovascular function in individuals with SCI ≥ T6.
2. Assess the effect of long-term tSCS on autonomic function in the subacute SCI phase: We will investigate the efficacy of long-term (total 18 sessions) tSCS on cardiovascular and pelvic organ functions.
3. Evaluate the sustained effect of tSCS on autonomic recovery six months after the onset of SCI: We will assess the sustained effect of repeated tSCS sessions (18 sessions) on cardiovascular and pelvic organ functions at 6-month post-SCI.

Participants will:

* Receive either transcutaneous spinal cord stimulation or "sham" spinal cord stimulation while inpatient in the first 8 weeks (Part A).
* Those willing and able to come after discharge or after the 8 weeks will be asked to come back and complete additional tSCS for a total of 18 weeks (Part B), with a follow-up period of 6 months. All participants will receive tSCS during this outpatient follow-up portion of the study.
* During assessment visits the researchers will perform a variety of exams including a neurologic, cardiovascular, pulmonary, bladder and bowel, physical, and autonomic exam, and will ask questions about quality of life and functioning. Participants will be asked to complete a test of how well their bowels are functioning (colonic transit test) and an abdominal X-Ray.

Researchers will compare those who receive tSCS to those who receive sham stimulation to see if tSCS is an effective treatment for improving the body's autonomic functioning following recent-onset SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 21-65 years of age.
2. SCI (non-progressive) at or above the T6 spinal segment.
3. Admitted to inpatient rehabilitation units or discharged from inpatient rehabilitation units but within 4 months since the onset on injury.
4. American Spinal Injury Association Impairment Scale (AIS) A-D for SCI.
5. Have stable medical condition that would permit participation in testing activities.
6. Willing and able to comply with all clinic visits and study-related procedures.
7. Able to understand and complete study-related questionnaires in English.
8. Have no painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing.
9. Are not currently pregnant or not intending to become pregnant during participation in this study.
10. Are volunteering to be involved in this study.
11. Must provide informed consent.

Exclusion Criteria:

1. Have autoimmune etiology of spinal cord dysfunction/injury
2. Have history of additional neurologic disease, such as stroke, MS, etc.
3. Have rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
4. Are ventilator dependent.
5. Have clinically significant, unmanaged, depression, ongoing alcohol and/or drug abuse.
6. Use any medication or treatment that in the opinion of the investigators indicates that it is not in the best interest of the participant to participate in this study.
7. Have Intrathecal baclofen pump.
8. Have cardiovascular, respiratory, bladder, or renal disease unrelated to SCI or presence of hydronephrosis or presence of obstructive renal stones.
9. Have severe acute medical issue that in the investigators' judgement would adversely affect the participant's participation in the study. Examples include, but are not limited to acute urinary tract infections, pressure sores, or unstable diabetes.
10. Have pacemakers, stimulators, medication pumps in the trunk, deep brain stimulators, metallic devices in the head such as aneurysm clips/coils and stents, vagus nerve stimulators.
11. Are a member of the investigational team or his/her immediate family.
12. Have history of severe allergy (i.e. allergic reaction that could not be treated with antihistaminic medication)
13. Have malabsorption syndrome, primary hyperthyroidism, and/or hypogonadism.
14. Have a history of seizures.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in systolic Blood Pressure (BP) | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  Continuous beat-by-beat BP will be measured using a finger photoplethysmography. This will be done throughout the study, including during orthostatic challenge using sit-up test.
Heart Rate (HR) monitoring during tSCS | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  Electrocardiography (ECG) at resting and during sit-up test
frequency and severity of uncontrolled BP episodes such as OH and autonomic dysreflexia (AD) in 24 hours. | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  24-hour BP monitoring obtained throughout the study using Finapres NOVA

SECONDARY OUTCOMES:
International Standards to document remaining Autonomic Function after Spinal Cord Injury (ISAFSCI) | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  Scores for questions on the ISAFSCI range from 0 to 2, with 0 representing complete loss of control and 2 representing normal functioning. Lower scores equal worse health functioning.
International Standards for Neurological Classification of Spinal Cord Injury | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  level and severity of damage to motor and sensory pathways will be determined by trained clinicians. Pin prick and light touch will be done by researchers on participant's left and right side. Check marks are given for each prick or touch that is felt by the participant, then tallied. Scores range from 0-56 for both the Left and Right side of the body, and 0-112 for the total score. High scores represent greater sensory functioning.
Autonomic dysfunction following Spinal Cord Injury (ADFSCI) measure | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  The Autonomic Dysfunction following SCI (ADFSCI) measure will be used to assess severity and frequency of autonomic dysreflexia. Greater scores equal greater frequency of autonomic dysfunction, ranging from 0 (never) to 4 (very often) for each item.
Numeric Pain Rating Scale | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  The Numeric Pain Rating Scale is a self-report measure, asking patients to circle a number on a scale ranging from 0 (no pain) to 10 (worst pain possible). Higher scores represent greater pain.
International SCI Pain Basic Dataset | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  Standardized questionnaire for the collection and reporting of pain in the SCI population. Scores range from 0 to 10, with higher scores indicating greater pain interference and worse functioning.
Neurogenic Bladder Symptom Score | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  The Neurogenic Bladder Symptom Score is a data collection form for measuring symptom burden of lower urinary tract functioning among those living with SCI. The Neurogenic Bladder Symptom Score (NBSS) is a validated 24 item questionnaire that measures bladder symptoms across 3 different domains: incontinence (scored 0-29), storage and voiding (scored 0-22), and consequences (scored 0-23); there is a single general urinary QOL question scored from 0 (pleased) to 4 (unhappy) [6]. For all domains, a higher score represents a worse symptom burden or QOL.
International SCI Lower Urinary Tract Function Basic Data Set (ISNCSCI) | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  The International SCI Lower Urinary Tract Function Dataset is a data collection form for the collection and reporting of lower urinary tract function in the SCI population. Participants are asked to mark either main or supplementary for type of bladder emptying, and then answer yes or no questions regarding type of appliances used to collect urinary incontinence, drugs with possible influence on urinary tract within the past 4 weeks, and any surgical procedures on the urinary tract. This data collection form does not use numbers and instead collects qualitative data only; there is no score range.
International SCI Bowel Function Basic Data Set (ISCIBFDS) | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  Standardized data collection form for the collection and reporting of bowel function in the SCI population. The International SCI Bowel Function Dataset is a data collection instrument that asks participants qualitative questions which are assigned a score. Select items are then totaled to compute the Neurogenic Bowel Dysfunction (NBD) score. Scores range from 0 to 14 or more, with higher scores indicating greater neurogenic bowel dysfunction.
Colonic Transit Time | Repeated measurements at baseline, post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at these 3 timepoints over 6 months.
  GI and colonic transit time will be assessed using radiopaque marker intake and an abdominal X-ray. Participants will take radiopaque markers for 6 days. On the 6th day, an abdominal X-ray will be taken. The movement of the radiopaque markers through the GI system will indicate colonic transit time, with slower transit time indicating possible neurogenic bowel.
Changes in Lower Urinary Tract and Bowel Function | Post-intervention (at time of discharge from inpatient rehabilitation), and 6 months post-spinal cord injury; assessed at 2 timepoints over 6 months.
  Maximum cystometric capacity measured via urodynamics. If appointments are available, participants will complete a urodynamic assessment in accordance with Good Urodynamic Practices recommended by the International Continence Society and international SCI Urodynamic data. Urodynamic assessments valuate how well the lower urinary tract, which includes the bladder, urethra, and sphincters, works to store and release urine. UDSs can help diagnose issues with the lower urinary tract and can show why there might be blockages or leaks. Abnormalities on the urodynamic assessment results may indicate neurogenic bladder.
Frequency and Severity of Adverse Events | Repeated measures at every study visit, over a period of 6 months.
  Serious Adverse Events and Adverse Events will be documented by study staff. For the purpose of this study, an adverse event (AE) is any untoward medical occurrence in a subject during participation in the clinical study or with use of the experimental agent being studied. An adverse finding can include a sign, symptom, abnormal assessment (vital signs, skin changes, neurological changes), or any combination of these.
  A serious adverse event (SAE) is any adverse event that results in one or more of the following outcomes:
  * Death
  * A life-threatening event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant disability/incapacity
  * A congenital anomaly or birth defect
  * An important medical event based upon appropriate medical judgment

CONTACTS AND LOCATIONS:
Overall Officials: Soshi Samejima, DPT, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States